CLINICAL TRIAL: NCT06957756
Title: Pharmacokinetics, Safety and Tolerability of BI 1584862 in Male and Female Participants With Different Degrees of Hepatic Impairment (Child-Pugh Class A, B, and C) Compared With Matched Male and Female Participants With Normal Hepatic Function (an Open-label, Non-randomized, Single-dose, Parallel, Individual-matched Design Trial)
Brief Title: A Study to Test How BI 1584862 is Taken up in the Blood of People With and Without Liver Problems
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1484-0009
Record Dates: First submitted 2025-05-02; First posted 2025-05-04 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Participants with mild hepatic impairment (Child-Pugh A) (Experimental)
  Interventions: Drug: BI 1584862
- Participants with moderate hepatic impairment (Child-Pugh B) (Experimental)
  Interventions: Drug: BI 1584862
- Participants with severe hepatic impairment (Child-Pugh C) (Experimental)
  Interventions: Drug: BI 1584862
- Participants with normal hepatic function (Experimental)
  Interventions: Drug: BI 1584862

INTERVENTIONS:
Drug: BI 1584862 — BI 1584862

SUMMARY:
This study is open to adults between 18 and 80 years of age. People with a body mass index (BMI) between 18 and 42 kg/m2 can take part. This study includes people with mild, moderate, and severe liver problems, and people without liver problems as a matching control. The purpose of this study is to find out how mild, moderate, and severe liver problems affect how the body handles a medicine called BI 1584862.

Participants take BI 1584862 once. Participants with liver problems are treated in a step-by-step approach with a few days in between for the doctors to review the data and to make sure the participants can tolerate the treatment. Participants may continue their regular treatment for their liver problems during the study.

Participants are in the study for about 5 weeks. During this time, they visit the study site 3 times. This also includes an overnight stay for 4 nights. During study visits, the doctors regularly check participants' health and take note of any unwanted effects. To assess the study endpoints, the site staff regularly takes blood samples.

ELIGIBILITY:
Inclusion criteria:

Inclusion criteria applicable to all participants

* Male or female participants
* Age of 18 to 80 years (inclusive)
* Body mass index (BMI) of 18.0 to 42 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Men participants must be willing and able to use contraception (condom, abstinence) from time point of administration of trial medication until 3 days after drug administration to prevent pregnancy and/or exposure of an existing embryo or fetus to the investigational product. Female partners do not need to use contraception
* Women of childbearing potential are allowed to participate provided they use a highly effective contraception from at least 30 days before the administration of trial medication until 30 days after administration of trial medication. The following methods of contraception are considered adequate for female participants of childbearing potential:

  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
  * Sexually abstinent (true abstinence, in line with the preferred and usual lifestyle of the subject)
  * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant.

Female participants are not considered to be of childbearing potential if they are either surgically sterilised (including hysterectomy) or postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of Follicle stimulating hormone (FSH) above 40 U/L and oestradiol below 30 ng/L is confirmatory).

Further inclusion criteria apply.

Exclusion criteria:

Exclusion criteria for all participants

* Any medical condition or finding in the medical examination (including blood pressure (BP), pulse rate (PR) or Electrocardiogram (ECG)) assessed as clinically relevant by the investigator (apart from any hepatic impairment and associated underlying diseases)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance (apart from values due to underlying disease)
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator (apart from underlying disease)
* For diabetics only: uncontrolled diabetes mellitus with an Hemoglobin A1c (HbA1c) > 9
* Severe gastrointestinal, renal (Estimated glomerular filtration rate (eGFR) Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) <40 ml/min/1.73 m2 for the hepatic impaired patients and eGFR CKD-EPI <90 ml/min/1.73 m2 for matched controls), respiratory, cardiovascular, metabolic, immunological or hormonal disorders assessed as clinically relevant by the Investigator.
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, repetitive fainting spells, or repetitive blackouts
* Relevant chronic or acute infections Further exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 4 days
Maximum measured concentration of the analyte in plasma (Cmax) | up to 4 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 4 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Arizona Clinical Trials, Chandler, Arizona
  - Omega Research Orlando, LLC, Orlando, Florida
  - American Research Corporation, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com